CLINICAL TRIAL: NCT00093808
Title: Phase II Study of Capecitabine in Combination With Vinorelbine and Trastuzumab for the First- or Second-LineTreatment of HER2+ Metastatic Breast Cancer
Brief Title: Capecitabine, Vinorelbine, and Trastuzumab in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0337; NCI-2012-02625 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000390344 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Trastuzumab; Capecitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- capecitabine + vinorelbine + trastuzumab (Experimental): Patients receive oral capecitabine twice daily on days 1-14, vinorelbine IV over 6-10 minutes on days 1 and 8, and trastuzumab (Herceptin^®) IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 3 months until disease progression and then every 6 months for up to 5 years.
  Interventions: Biological: trastuzumab; Drug: capecitabine; Drug: vinorelbine tartrate

INTERVENTIONS:
Biological: trastuzumab
Drug: capecitabine
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and vinorelbine, work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor killing substances to them without harming normal cells. Giving capecitabine and vinorelbine together with trastuzumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving capecitabine and vinorelbine together with trastuzumab works in treating patients who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall response rate in patients with HER2/neu-overexpressing metastatic breast cancer treated with first- or second-line therapy comprising capecitabine, vinorelbine, and trastuzumab (Herceptin^®).

Secondary

* Determine the time to disease progression, duration of response, and overall survival of patients treated with this regimen.
* Determine the safety profile of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral capecitabine twice daily on days 1-14, vinorelbine IV over 6-10 minutes on days 1 and 8, and trastuzumab (Herceptin^®) IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until disease progression and then every 6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed invasive breast cancer

  * Metastatic disease
* HER2/neu-positive by immunohistochemistry (3+ by HercepTest^™ or equivalent) OR positive for amplification by fluorescent in situ hybridization

  * Testing may be performed in the primary tumor or the metastatic site
* Received prior anthracycline or taxane as adjuvant therapy or for metastatic disease
* Measurable disease

  * At least one measurable lesion ≥ 2.0 cm by CT scan or MRI OR ≥ 1.0 cm by spiral CT scan
  * The following are considered non-measurable disease:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* No bone metastases as the only evidence of metastasis
* Previously treated CNS metastases allowed provided disease has been stable for ≥ the past 3 months
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female or male

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 100,000/mm^3
* No known uncontrolled coagulopathy

Hepatic

* Bilirubin ≤ 3.0 times the upper limit of normal (ULN)
* One of the following must be true:

  * AST or ALT ≤ 5 times ULN AND alkaline phosphatase normal
  * Alkaline phosphatase ≤ 5 times ULN AND AST or ALT normal
  * Alkaline phosphatase ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
* INR ≤ 1.5 times ULN

Renal

* Calcium ≤ 11.5 mg/dL
* Creatinine ≤ 1.5 times ULN
* Creatinine clearance ≥ 30 mL/min

Cardiovascular

* LVEF ≥ 50% by MUGA or echocardiogram
* No clinically significant (i.e., active) cardiac disease
* No congestive heart failure
* No symptomatic coronary artery disease
* No myocardial infarction within the past 12 months
* No cardiac arrhythmia not controlled with medication

Gastrointestinal

* Able to take oral medication
* No lack of physical integrity of the upper gastrointestinal tract
* No clinically significant malabsorption syndrome

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after study participation
* No history of allergy or hypersensitivity to study drugs, drug product excipients, including polysorbate 80, or chemically similar agents
* No prior unanticipated severe reaction to fluoropyrimidine therapy
* No know hypersensitivity to fluorouracil
* No known dihydropyrimidine dehydrogenase deficiency
* No history of uncontrolled seizures or CNS disorders
* No clinically significant psychiatric disability that would preclude giving informed consent or study compliance
* No other serious uncontrolled infection or disease
* No other malignancy within the past 5 years except cured basal cell skin cancer, carcinoma in situ of the cervix, or contralateral breast cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior adjuvant trastuzumab (Herceptin^®) allowed as adjuvant or first-line therapy for metastatic disease
* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* No more than 1 prior chemotherapy regimen in the advanced or metastatic (non-adjuvant) setting
* No prior continuous (≥ 24 hours) fluorouracil infusion
* No prior capecitabine
* No prior oral fluoropyrimidines (e.g., eniluracil and fluorouracil, uracil and tegafur, S1, or emitefur)

Endocrine therapy

* At least 1 day since prior hormonal therapy
* No concurrent hormonal therapy

Radiotherapy

* More than 4 weeks since prior radiotherapy to the axial skeleton (i.e., skull, spinal column, sternum, or ribs)
* No concurrent radiotherapy

Surgery

* More than 4 weeks since prior major surgery
* No prior organ allografts requiring immunosuppressive therapy

Other

* More than 4 weeks since prior investigational drugs
* No concurrent sorivudine or its chemically related analogues (e.g., brivudine)
* No concurrent allopurinol, metronidazole, or cimetidine
* No other concurrent cytotoxic agents
* No other concurrent investigational drugs
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-08; Primary Completion 2008-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Winston Tan, MD, FACP, Study Chair — Mayo Clinic
Locations (147):
- United States (147):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Result] Tan WW, Allred JB, Salim M, Flynn P, Fishkin PA, Stella PJ, Wiesenfeld M, Bernath AM, Fitch TR, Perez EA. Phase II interventional study (N0337) of capecitabine in combination with vinorelbine and trastuzumab for first- or second-line treatment of HER2-positive metastatic breast cancer: a north central cancer treatment group trial. Clin Breast Cancer. 2012 Apr;12(2):81-6. doi: 10.1016/j.clbc.2012.01.001. PMID 22444716
- [Derived] Chumsri S, Sperinde J, Liu H, Gligorov J, Spano JP, Antoine M, Moreno Aspitia A, Tan W, Winslow J, Petropoulos CJ, Chenna A, Bates M, Weidler JM, Huang W, Dueck A, Perez EA. High p95HER2/HER2 Ratio Associated With Poor Outcome in Trastuzumab-Treated HER2-Positive Metastatic Breast Cancer NCCTG N0337 and NCCTG 98-32-52 (Alliance). Clin Cancer Res. 2018 Jul 1;24(13):3053-3058. doi: 10.1158/1078-0432.CCR-17-1864. Epub 2018 Mar 12. PMID 29530935

RESULTS

PARTICIPANT FLOW:
Groups:
- Capecitabine + Vinorelbine + Trastuzumab: Treatment followed a 21-day cycle. Capecitabine was administered orally twice daily at a dose of 825 mg/m^2 on days 1 to 14, vinorelbine was administered intravenously (IV) at a dose of 25 mg/m^2 on days 1 and 8 every 3 weeks, and trastuzumab was administered IV at a dose of 6 mg/kg on day 1 of every 3-week cycle (except cycle 1, when patients were given a loading dose of 8 mg/kg).
Period: Overall Study
Arm/Group | Capecitabine + Vinorelbine + Trastuzumab
Started | 47
Completed | 45
Not Completed | 2
Not completed — Cancel participation before receiving tx | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Patients who completed the study or deemed a protocol violation were included in all analyses unless otherwise specified.
Arm/Group | Capecitabine + Vinorelbine + Trastuzumab
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Response Rate
Description: A confirmed tumor response is defined to be either a Complete Response (CR) or Partial Response (PR) noted as the objective status on 2 consecutive evaluations at least 6 weeks apart. All patients meeting the eligibility criteria who have signed a consent form and initiated study medication will be evaluable for response. The proportion of confirmed tumor responses will be estimated by the number of tumor regressions that meet the RECIST criteria for a confirmed CR or PR divided by the total number of evaluable patients. A 95% confidence interval for the true confirmed response rate will be calculated using the properties of the binomial distribution. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 5 years
Population: Patients who completed the study were included in all analyses unless otherwise specified.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Capecitabine + Vinorelbine + Trastuzumab
Number analyzed (Participants) | 45
proportion of patients | 0.67 [0.51 to 0.80]

2. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression is defined as the time from registration to disease progression. Patients who died without documentation of progression will be considered to have progressed on the date of their death. If a patient starts treatment and fails to return for any evaluations, that patient will be censored for progression of disease at day one post-registration. Otherwise, for patients that do not progress, censoring will occur at the last follow up date. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as at least a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions or unequivocal progression of existing non-target lesions.
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine + Vinorelbine + Trastuzumab
Number analyzed (Participants) | 46
months | 11.3 [8.4 to 16.7]

3. Secondary Outcome: Duration of Response as Measured by RECIST Criteria
Description: Duration of response is defined for all eligible patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a Complete Response (CR) or Partial Response (PR) to the date progression is documented. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine + Vinorelbine + Trastuzumab
Number analyzed (Participants) | 46
months | 13.2 [8.6 to 23.2]

4. Secondary Outcome: Overall Survival as Assessed by Time
Description: Overall survival: The overall survival or survival time is defined as the time from registration to death due to any cause. The distribution of overall survival will be estimated using the method of Kaplan-Meier method.
Time Frame: Up to 5 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine + Vinorelbine + Trastuzumab
Number analyzed (Participants) | 46
months | 28.5 [24.8 to 36.4]

ADVERSE EVENTS:
Time Frame: Adverse events are collected 2 weeks prior to registration, at each evaluation , and at end of treatment during the Active-Monitoring Phase; up to 5 years post registration.
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized until June 30, 2011. CTCAE version 4.0 will be utilized for expedited adverse event reporting only, beginning July 1, 2011. Adverse events data collected for patients who received and completed at least one cycle of treatment are reported below (i.e. for patients who completed the study or deemed a protocol violation).
Arm/Group | Capecitabine + Vinorelbine + Trastuzumab
Serious Adverse Events (participants affected / at risk) | 9/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine + Vinorelbine + Trastuzumab (N=46)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine + Vinorelbine + Trastuzumab (N=46)
Hemoglobin decreased (Blood and lymphatic system disorders) | 11 (23)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 2 (2)
Cataract (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 2 (9)
Abdominal pain (Gastrointestinal disorders) | 5 (9)
Constipation (Gastrointestinal disorders) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 30 (113)
Dyspepsia (Gastrointestinal disorders) | 3 (4)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 8 (10)
Nausea (Gastrointestinal disorders) | 8 (9)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (8)
Chest pain (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 45 (356)
Fever (General disorders) | 1 (1)
Injection site reaction (General disorders) | 6 (19)
Visceral edema (General disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (3)
Bladder infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Lip infection (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (5)
Creatinine increased (Investigations) | 9 (13)
INR increased (Investigations) | 1 (2)
Leukocyte count decreased (Investigations) | 11 (32)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 39 (196)
Platelet count decreased (Investigations) | 8 (38)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 6 (8)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (7)
Dehydration (Metabolism and nutrition disorders) | 4 (5)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (5)
Serum potassium decreased (Metabolism and nutrition disorders) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 25 (136)
Fibrosis (Musculoskeletal and connective tissue disorders) | 2 (8)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 27 (139)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 2 (8)
Headache (Nervous system disorders) | 3 (7)
Neuralgia (Nervous system disorders) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 9 (23)
Peripheral sensory neuropathy (Nervous system disorders) | 32 (298)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (9)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (12)
Proteinuria (Renal and urinary disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (20)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 25 (202)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 11 (31)
Hot flashes (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Lymphedema (Vascular disorders) | 1 (3)
Thrombosis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes